CLINICAL TRIAL: NCT03437135
Title: Screening and Characterization of Hearing Disorders in Diabetic Persons.
Acronym: DeCaTAuDiab
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-371
Record Dates: First submitted 2018-01-12; First posted 2018-02-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2018-02

CONDITIONS: Diabetes; Hearing Problems
Keywords: diabetes; hearing problems; otoscopy
MeSH Terms: conditions — Diabetes Mellitus; Hearing Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Witness patients: Healthy Volunteers
  Interventions: Diagnostic Test: Glasgow Hearing Status Inventory questionnaire
- Type 1 diabetic patients: patients with type 1 diabetes
  Interventions: Diagnostic Test: Glasgow Hearing Status Inventory questionnaire
- Type 2 diabetic patients: patients with type 2 diabetes
  Interventions: Diagnostic Test: Glasgow Hearing Status Inventory questionnaire

INTERVENTIONS:
Diagnostic Test: Glasgow Hearing Status Inventory questionnaire — This is a questionnaire of the hearing quality presenting eleven questions. This is allows to determine the quality of the hearing status of the patients. It is enough to answer the various questions "yes" or "no".

SUMMARY:
Diabetes is now the most common chronic disease, affecting nearly 6% of the population in Western populations. Diabetic neuropathy is a priori the most common and the most common specific complications of diabetes. It can of course touch the lower limbs, the vegetative nervous system as well as the cranial nerves. However, the association between hearing impairment and diabetes has always been controversial on the basis of conflicting literature data. Are auditory disorders an underestimated complication of diabetes? A meta-analysis made in 2013, examined the scientific literature between 1950 and 2011 and of the 3158 citations, only 13 articles were selected. This study found that hearing impairment in diabetic patients was 2.1 times more prevalent than in non-diabetic matched subjects. In addition, the age / aging factor is associated with the prevalence of hearing loss and diabetes. However, it also appears that the link between diabetes and hearing impairment is more pronounced among young people than older people. In order to document the influence of diabetic pathology on hearing, Investigator have set up a search audiological exploration platform within the department of Endocrinology-Diabetology of Clermont-Ferrand University Hospital. It will be proposed a hearing screening (duration 30 minutes) and a questionnaire to diabetic patients of the service. In the context of a positive screening, that is to say that one of the tests carried out reveals the presence of a hearing disorder, an in-depth assessment of the hearing will be carried out to better characterize the origin of the auditory disturbance (duration 60-90 minutes). These different tests are based on the listening of sounds requiring or not the participation of patient. Thus, the results of the various tests will make it possible to classify the impairment of hearing in (1) peripheral impairment (dysfunction of certain cells of your ear involved in the amplification of sounds), and / or (2) in neural damage (dysfunction of your auditory nerve).

DETAILED DESCRIPTION:
Diabetes is now the most common chronic disease since it affects western populations such as France almost 6% of the population. This disease is particularly costly for social protection systems, not only for the cost of daily care but also by the occurrence of Chronic complications that are leading to major co-morbidities. Thus, diabetes is a major cardiovascular risk factor. Diabetes also leads to micro-angiopathic complications: Diabetic retinopathy eventually ends up in evolved forms to the first cause of young subject blindness in developed countries. Nephropathy is one of the first causes of terminal renal failure leading to extra renal treatment.

Diabetic neuropathy seems to be the most common and the most common of the specific complications of diabetes. It can of course touch the lower limbs, most often training a symmetrical and distal motor polyneuritis, responsible for the term of Neuro arthropathy of Charcot. The vegetative nervous system can also be achieved with cardiovascular, gastrointestinal, genitourinary, neuro-vascular, metabolic and pupil consequences. The injuries of the cranial nerves are also possible and are most frequently characterized by facial paralysis or motor eye nerves.

The association between hearing disorders and diabetes has always aroused controversy on the part of contradictory literature data. Are hearing disorders an underestimated complication of diabetes? A recent meta-analysis of 2013, examined the scientific literature between 1950 and 2011 and of the 3158 citations, only 13 articles were selected (with more than 20 000 participants). This study found that hearing disorders in diabetic patients were 2.1 times more prevalent than in non-diabetic paired subjects. In addition, the age/aging factor is associated with the prevalence of hearing impairment and diabetes. However, it also appears that the link between diabetes and hearing disorder is more pronounced among young people than the elderly.

Nevertheless, it is regrettable that in the majority of the "diabetes-hearing disorders" studies were not exhaustive from the point of view of the documentation of the alteration of the hearing function. Indeed, the indices of impairment of the hearing are essentially based on a review of the audiograms. No more relevant objective test, allowing to evaluate more precisely the different functional compartments of the inner ear, has been achieved. Indeed, it would be wise to elucidate which (s) are the targets (s) of the diabetes. Classical hearing impairment mainly affects cochlear sensory cells and more specifically external hair cells. However, it is possible to envisage that the alteration of the micro-vascularization of the vascular Streak (ischemic disorders), a selective expectation of the nerve fibers (hearing neuropathy), the metabolic disturbances at the mitochondrial level, Oxidative stress with free radical production, advanced glycation products (AGE, advanced glycation end-products).

Objectives:

* The primary objective is the assessment of the prevalence of hearing impairment (with or without clinical manifestation) in a population of type 1 and type 2 diabetic persons treated and followed during a hospitalization or consultation in the Department of Endocrinology-Diabetology of the CHU de Clermont-Ferrand.
* The second objectives are:

Identify the proportion of patients with a peripheral explanation for their hearing impairment (involvement of the outer ciliated cells, 'classic deafness) Identify the proportion of patients who have a neural explanation for their hearing impairment (hearing-type neuropathy) And categorize types of hearing impairment by types of diabetes, its balance, age, absence or absence of complication, age of patient, sex of patient, noise exposure in a professional manner or as a part of recreation, taking ototoxic drugs, smoking.

ELIGIBILITY:
Inclusion Criteria:

* type 1 or type 2 diabetic patients

Exclusion Criteria:

* history of otological surgical act
* presence of neurological or psychiatric disorders that may impair the quality of explorations
* presence of a obstructive wax stopper or au foreign body found in the simple otoscopy (or impossibility of this extraction).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetic persons
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
presence or not of an ear wax cap | At day 1 (during the inclusion and screening consultation)
  A single ostoscopie is performed using a portable otoscope and single-use Speculum to verify the absence of any wax cap.

SECONDARY OUTCOMES:
mobility of the eardrum-ossicular | At day 1 (during the inclusion and screening consultation)
  From a tympanometry probe with a single-use mouthpiece, the mobility of the eardrum is studied and therefore the functional state of the middle ear.
Study of Stapedius reflex | At day 1 (during the inclusion and screening consultation)
  From a tympanometry probe with a single-use mouthpiece, the study of Stapedius reflex allows to evaluate the functionality of a reflex neurological loop of the brainstem. The stapedium reflex rating is "present " or "absent "
Study of acoustic ear emissions | At day 1 (during the inclusion and screening consultation)
  A measuring probe is carefully inserted into the external ear canal and an analysis of the overall responses of the cochlea is carried out following the application of an acoustic stimulation. The ear emission rating is "present " or "absent
the auditory threshold | At day 1 (during the inclusion and screening consultation)
  A tonal audiogram for 6 frequencies from 250 to 8000 will be achieved to determine of auditory threshold
the functionality of external ciliated cells (ECC) | At day 2 (during the exploration consultation)
  this is a non-invasive, simple, fast and objective assay for exploring the functionality of external ciliated cells (ECC). This test is similar test in some aspects to the test of acoustic ear emissions, but allows to have an analysis of cochlear answers (and more specifically ECC) not global but between 1000 hertz and 8000 hertz
Early auditory evoked potentials (or eAEP) | At day 2 (during the exploration consultation)
  Electrodes are positioned at specific points at the level of the scalp (according to the system 10/20, at the level of the vertex and in frontal-median Fp).
frequency selectivity of the patient | At day 2 (during the exploration consultation)
  the objective of this test is to measure the selectivity in frequency for three frequencies (1000, 2000 and 4000hertz).

CONTACTS AND LOCATIONS:
Overall Officials: Igor TAUVERON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France